CLINICAL TRIAL: NCT04793516
Title: Development of a Virtual Reality Spatial Retraining Therapy to Improve Neglect in Stroke Survivors
Acronym: VR-SRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Peii Chen, Senior Research Scientist, PI, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-996-17
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Spatial Neglect
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-based spatial retraining (Experimental): Game-like therapy activities will be taken place in a virtual environment, provided through an immersive head-mounted display.
  Interventions: Other: VR Therapy Game

INTERVENTIONS:
Other: VR Therapy Game — Participants will complete 15 sessions of VR-based therapy modules developed for use in helping people with spatial neglect. These 15 sessions will be completed over 4-5 weeks.

SUMMARY:
Participants in this study will help test and develop a virtual reality (VR) system that is being designed to help people with spatial neglect after stroke.

DETAILED DESCRIPTION:
Participants in this study will be tested to see if they have spatial neglect after their stroke, and the severity of such. Spatial neglect is a disorder that may occur after a stroke that leads to a person paying more attention to one side of their body over the other. Each testing session, they will perform paper and pencil neglect tests before and after playing a VR video game that is being designed as a potential future treatment. They will also give feedback on the game after the session is over. People who have spatial neglect after stroke are encouraged to apply.

ELIGIBILITY:
Inclusion Criteria:

* Read and speak English fluently
* Have a history of one stroke event that injured one cerebral hemisphere
* Presence of moderate to severe spatial neglect

Exclusion Criteria:

* History of progressive neurological disorders
* History of significant psychiatric disorders
* History of vestibular disorders
* Living outside a 50-mile radius of Kessler Foundation (located in West Orange, NJ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral Inattention Test | At baseline, after intervention, and two weeks after intervention
  A battery of visuospatial tests using paper and pencil to perform line crossing, star cancellation, letter cancellation, line bisection, figure copying, and drawing. The test is scored from 0 to 146, with higher values indicating better performance.

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire | After intervention
  A 16-item questionnaire asking for adverse feelings related to the virtual reality experience. Example items are eye strain, difficulty concentrating, headache, and burping. Each item is rated none, slight. moderate, or severe.
Semi-structured interview | Two weeks after intervention
  A 10-minute phone interview will be conducted to explore the subjective experience of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peii Chen, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT04793516/ICF_000.pdf